CLINICAL TRIAL: NCT00149448
Title: Effectiveness of the TB Contact Priority Model
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1304
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

INTERVENTIONS:
Behavioral: TB Contact Priority Model

SUMMARY:
The broad purpose of this project, proposed by investigators at the University of Alabama at Birmingham and the State of Alabama Department of Public Health, is to use a behaviorally focused education that has been proven effective to enhance the accuracy and efficiency of the contact investigation process. The behaviorally focused intervention will focus on enabling public health workers to understand and implement a recently published model of TB transmission.

DETAILED DESCRIPTION:
BACKGROUND:

Investigation of contacts of patients with active pulmonary tuberculosis (TB) is an important epidemiological tool in TB control. Unfortunately, due to budgetary and resource constraints, many health departments struggle to fulfill their responsibility of TB control through contact investigation.

DESIGN NARRATIVE:

Primary outcome The primary outcome of this project is to examine the clinical effectiveness of the TB transmission model. This will be done by examining the sensitivity and specificity of the model when used in a field application.

Key secondary outcomes Evaluation of the efficiency of contact investigation (two outcomes: 1) weekly average time to tuberculin skin test placement for high risk contacts, 2) weekly average time to the close of the contact investigation.) Qualitative assessment of individuals who are incorrectly predicted by the model to have a negative tuberculin skin test

ELIGIBILITY:
B field workers for the Alabama Department of Public Health.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)